CLINICAL TRIAL: NCT03724409
Title: Selective Intra-arterial Injection of Peptide Receptor Radionuclide Therapy (PRRT) in Neuroendocrine Tumor Patients With Liver Metastases
Brief Title: Selective Intra-arterial Injection of PRRT in Neuroendocrine Tumor Patients With Liver Metastases
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Pandemic
Sponsor: Sandeep Laroia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sandeep Laroia, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201805910; P50CA174521 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Neuroendocrine Tumors
Keywords: PRRT; Radionuclide; DOTATOC; intra-arterial; peptide receptor radiotherapy
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 90Y-octreotide, DOTA-Tyr(3)-

STUDY DESIGN:
Intervention Model Description: This is a sequential early phase 1 study using Storer's phase 1 design B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Subject will be administered 2.96 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC
- Cohort 2 (Experimental): Subject will be administered 3.33 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC
- Cohort 3 (Experimental): Subject will be administered 3.7 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC
- Cohort 4 (Experimental): Subject will be administered 4.17 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC
- Cohort 5 (Experimental): Subject will be administered 4.44 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC
- Cohort 6 (Experimental): Subject will be administered 5.18 gigabecquerels of [90]Y-DOTATOC intra-aterially to the liver
  Interventions: Drug: [90]Y-DOTATOC

INTERVENTIONS:
Drug: [90]Y-DOTATOC — Intra-arterial infusion to the liver of [90]Y-DOTATOC. The administered dose is determined by cohort and is dependent upon the results of the previous cohort.
  Other Names: 90Y-DOTATOC; 90Y-DOTA-Phe1-tyr3-Octreotide; [90]Yttrium-DOTATOC

SUMMARY:
This is a safety study to determine the phase 1 starting dose of [90]Yttrium-DOTATOC when it is administered intravenously for patients with neuroendocrine tumors that have spread to the liver.

DETAILED DESCRIPTION:
[90]Yttrium-DOTATOC is a radioactive drug used for peptide receptor radionuclide therapy (PRRT). In other studies, 90Y-DOTATOC has been administered through a vein (IV) to target somatostatin receptor positive tumor tissue. The DOTATOC identifies the tumor through the somatostatin receptor and links to it, attaching the radioactive molecule 90Yttrium to the malignant cell.

This study expands the initial work to examine if administering the drug 90Y-DOTATOC directly to the liver is safe for patients with neuroendocrine tumors whose disease has spread to their tumor. We don't know how of the 90Y-DOTATOC is safe to administer. We want to learn what the maximum safe dose is and what the side effects are related to that dose.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to provide informed consent
* Pathologically well-differentiated neuroendocrine tumor (i.e. grade 1 or grade 2).
* Primary tumor location should be known or believed to be midgut.
* At least one tumor in the liver that is positive with [68]Ga-DOTATATE (NETSPOT). Imaging must be performed within the past 6 months.
* Liver lesions not amendable to other therapies (surgery, ablation) and have progressed after treatment with octreotide/lanreotide and/or other treatments. (everolimus, sunitinib).
* Karnofsky performance status of at least 70
* Absolute neutrophil count of at least 1,000 cells/mm3
* Platelet count of at least 90,000 cells / mm3
* Total bilirubin ≤ 2 x the upper limit of normal when adjusted for age
* AST and ALT ≤ 5 x the upper limit of normal when adjusted for age
* Serum creatinine ≤ 1.2 mg/dl; if serum creatinine is >1.2 mg/dl nuclear GFR will used for potentially eligible participants.
* Agrees to contraception.

Exclusion criteria:

* Liver tumor involvement greater than 70% by cross sectional imaging
* Extra-hepatic visceral and osseous metastases
* Concomitant therapy for tumor (except for somatostatin analogs or bisphosphonates)
* Previous PRRT or other liver directed therapy within 12 months of consent
* Women who are pregnant, breast feeding or breast pumping.
* Another concurrent malignancy on active therapy
* Previous external-beam radiation therapy to a kidney (including scatter dose)
* Therapeutic investigational drug within 4 weeks of therapy.
* Subjects for whom, in the opinion of their physician, a 24-hour discontinuation of somatostatin analogue therapy represents a health risk.
* Sandostatin LAR injection within 4 weeks or lanreotide injection within 8 weeks of proposed therapy.
* Inability to lie down supine for study procedure.
* Reaction to IV contrast used for the angiogram.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring hospitalization, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Change in liver enzymes | Through 6 weeks after treatment
  Evaluate liver toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) severity scale for liver enzymes
Change in platelet counts | Through 6 weeks after treatment
  Evaluate bone marrow toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) severity scale for platelet count
Change in absolute neutrophil count | Through 6 weeks after treatment
  Evaluate bone marrow toxicity using using the Common Terminology Criteria for Adverse Events (CTCAE) severity scale for absolute neutrophil count

SECONDARY OUTCOMES:
90Y-DOTATOC distribution | 48h post-infusion
  Determine the distribution of 90Y-DOTATOC using post-treatment imaging

CONTACTS AND LOCATIONS:
Overall Officials: M. S O'Dorisio, MD, PhD, Study Chair — University of Iowa; Sandeep Laroia, MD, Principal Investigator — University of Iowa
Locations (1):
- The Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as per approved IRB application and the subject's opt-in preferences. Data will not be provided from subjects who decline data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Considered upon request.
Access Criteria: Contact study PI regarding data sharing. A non-disclosure agreement may be required between institutions dependent upon the data requested.

REFERENCES:
- [Background] Kennedy A, Bester L, Salem R, Sharma RA, Parks RW, Ruszniewski P; NET-Liver-Metastases Consensus Conference. Role of hepatic intra-arterial therapies in metastatic neuroendocrine tumours (NET): guidelines from the NET-Liver-Metastases Consensus Conference. HPB (Oxford). 2015 Jan;17(1):29-37. doi: 10.1111/hpb.12326. Epub 2014 Sep 4. PMID 25186181